CLINICAL TRIAL: NCT06932926
Title: Remineralization Potential Of Egg Shell Hydrogel Versus Fluoride Varnish On Early Carious White Spot Lesions In Anterior Primary Teeth: A Randomized Controlled Trial
Brief Title: Remineralization Effect Of Egg Shell Versus Fluoride Varnish On Early Carious White Spot Lesions In Primary Teeth
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Bahr Hussein Youssef, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Faculty of dentistry CairoU
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Egg shell hydrogel. (Experimental)
  Interventions: Drug: Egg shell hydrogel
- Fluoride varnish. (Active Comparator): five percent sodium fluoride varnish (Charm varnish -Dentkist- Korea).
  Interventions: Drug: Fluoride varnish

INTERVENTIONS:
Drug: Egg shell hydrogel — I. Nano-eggshell powder preparation: After cleaning, A small crack will be made in each eggshell to split it into two halves to evacuate the content. The eggshells will be disinfected in a hot water at 100°C for 10 minutes to facilitate the detachment of the inner membrane. They will be exposed to steam sterilization. Then they will be crushed using a sterile mortar and pestle. The crushed particles will be milled using a zirconia ball-milling machine at 200 rpm . This will result in a nano-sized eggshell powder to incorporate them into a gel form.
  II. Preparation of eggshell hydrogel formulations: through dispersing a suitable concentration of egg shell powder in distilled water, followed by dissolving the gelling agent; sodium carboxymethyl cellulose at a concentration of 5-10% under continuous stirring. The formed hydrogel will be kept at 8°C for a period of 24 hours before further use. This will produce a paste of consistency that is appropriate for handling and application.
  Arms: Egg shell hydrogel.
Drug: Fluoride varnish — five percent sodium fluoride varnish (Charm varnish -Dentkist- Korea).
  Arms: Fluoride varnish.

SUMMARY:
The goal of this clinical trial is to to assess the remineralization potential of Egg shell hydrogel versus fluoride varnish in early carious white spot lesions in anterior primary teeth.

The main question it aims to answer is:What is the remineralization potential of egg shell hydrogel on early carious white spot lesions compared to fluoride varnish in anterior primary teeth? Researcher will compare egg shell hydrogel with fluoride varnish to see if it is able to promote lesion remineralization.

interventions that will be given to participasnts: egg shell hydrogel & five percent sodium fluoride varnish

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3 to 5 years, in good general health, and medically free.
2. Prescence of at least one WSL on anterior primary teeth with an ICDAS II score of one or two.
3. Cooperative patients who will comply with follow-ups.
4. Parents who accept to sign informed consent.

Exclusion Criteria:

1. Uncooperative children.
2. Children with a physical disability or medical disability.
3. Children with teeth that shows enamel hypoplasia.
4. Children that have received a fluoride supplement or professional topical fluoride application at least 3 months before the study.
5. Parents refuse to give written formed consent.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Remineralization potential. | at 6th , 18 and 30th week
  change in minerals content of the lesion , will be assessed using diagnodent scores ( minimum value is 0 and maximum value is 99 ) higher scores means worse outcome .

SECONDARY OUTCOMES:
Activity of the lesion | will be assessed using Nyvad's criteria at 6th , 18 and 30th week
  whether the lesion is active or in active , will be assessed using Nyvad's criteria ( minimum value is score 0 and maximum value is score 9) higher scores means worse outcome .
Oral hygiene | at 6th , 18 and 30th week
  Oral hygiene status will be assessed using modification of OHI-S ( Simplified Oral Hygiene Index ) minimum value is score 0 and maximum value is score 3 higher score means worse outcome .